CLINICAL TRIAL: NCT02718989
Title: Modulation of H-reflex After Application of Electric Currents in Healthy People. Effects on Myotonometer Properties.A Pilot Study
Brief Title: Modulation of H-reflex After Application of Electric Currents in Healthy People
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Castilla-La Mancha (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: ddsm25
Record Dates: First submitted 2016-03-03; First posted 2016-03-24 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Spasticity
Keywords: H-reflex; TENS; Tone
MeSH Terms: conditions — Muscle Spasticity | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 10 Kilohertz (KHz) (Experimental): Transcutaneous application of 10 Kilohertz (KHz) current over the back for a 40 minutes session. The intensity of the current will increase until participants report a "strong but comfortable" sensation, just below motor threshold.
  Interventions: Device: Transcutaneous Electrical Stimulation; Device: 10Kilohertz (KHz)
- Transcutaneous Electrical Stimulation (Experimental): Transcutaneous application of TENS current over the back for a 40 minutes session. The intensity of the current will increase until participants report a "strong but comfortable" sensation, just below motor threshold. Currents parameters are frequency 100 Hz and pulse width 100 microseconds
  Interventions: Device: Transcutaneous Electrical Stimulation
- Sham stimulation (Sham Comparator): Electrodes are placed over the back for a 40 minutes in the same manner as experimental groups, but will be applied a sham electrical stimulation increasing the current intensity of an unconnected channel.
  Interventions: Device: Sham stimulation

INTERVENTIONS:
Device: Transcutaneous Electrical Stimulation — TENS transcutaneous electrical stimulation over the back the electrotherapy device Myomed 932. (Enraf-Nonius, Delft, Netherlands)
  Other Names: TENS
  Arms: 10 Kilohertz (KHz); Transcutaneous Electrical Stimulation
Device: 10Kilohertz (KHz) — 10 KHz transcutaneous electrical stimulation over back through the electrotherapy device Myomed 932. (Enraf-Nonius, Delft, Netherlands)
  Arms: 10 Kilohertz (KHz)
Device: Sham stimulation — Sham transcutaneous electrical stimulation over back through the electrotherapy device Myomed 932. (Enraf-Nonius, Delft, Netherlands)
  Arms: Sham stimulation

SUMMARY:
The purpose of this study is to determinate whether the application of electric currents produce changes in the excitability of alpha moto neurone. Moreover evidence whether the effect of the electric currents can change the tone of the muscle under stimulation in healthy volunteers

DETAILED DESCRIPTION:
In the last years several experimental studies have evidenced that the transcutaneous electric nerve stimulation (TENS) in peripheric application can cause a decrease of spasticity and modulation of H-reflexes.

But if the application is in the central nervous system the results are different. So the purpose of this study is quantify the modulation of the excitability of alpha moto neurone when the application of the current is in the central nervous system compared with a sham group.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be volunteer healthy students of Physiotherapy, University of Castilla - La Mancha, older than 18 years.

Exclusion Criteria:

* Neuromuscular disease
* Epilepsy
* Trauma, surgery or pain affecting the upper limb, shoulder girdle or cervical area
* Osteosynthesis material in the upper limb
* Diabetes
* Cancer
* Cardiovascular disease
* Pacemaker or other implanted electrical device
* Take any drug (NSAIDs, corticosteroids, antidepressants, analgesics, antiepileptics, ...) during the study and in the previous 7 days.
* Presence of tattoos or other external agent introduced into the treatment or assessment area.
* Pregnancy
* Sensitivity disturbance in lower limb

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-06 (Estimated); Primary Completion 2017-08 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
Baseline H reflex | baseline at 0 min.
  H-reflex data are obtained by EMG signal. The EMG electrode (SignalConditioningElectrodes v2.3, Delsys Inc., USA) is fixed on triceps surae by the SENIAM protocol (www.seniam.org). The stimulator electrode is fixed on the peroneus nerve, in the popliteal fossa.
During treatment H reflex | During treatment at 33min.
  H-reflex data are obtained by EMG signal. The EMG electrode (SignalConditioningElectrodes v2.3, Delsys Inc., USA) is fixed on triceps surae by the SENIAM protocol (www.seniam.org). The stimulator electrode is fixed on the peroneus nerve, in the popliteal fossa.
Post treatment H reflex | Immediately after treatment at 40 min.
  H-reflex data are obtained by EMG signal. The EMG electrode (SignalConditioningElectrodes v2.3, Delsys Inc., USA) is fixed on triceps surae by the SENIAM protocol (www.seniam.org). The stimulator electrode is fixed on the peroneus nerve, in the popliteal fossa.

SECONDARY OUTCOMES:
Baseline muscle tone | Baseline at 0 min.
  This outcome measure is obtained by a device named MyotonPro. It is a commercial device made to calculate myotonometrics properties of the muscle. It is a non-invasive method to calculate the muscle tone. The investigators obtained many parameters like muscle stiffness, frequency and decrement.
Muscle tone during treatment | During treatment at 35 min.
  This outcome measure is obtained by a device named MyotonPro. It is a commercial device made to calculate myotonometrics properties of the muscle. It is a non-invasive method to calculate the muscle tone. The investigators obtained many parameters like muscle stiffness, frequency and decrement.
Muscle tone post-treatment | Post-treatment at 42min
  This outcome measure is obtained by a device named MyotonPro. It is a commercial device made to calculate myotonometrics properties of the muscle. It is a non-invasive method to calculate the muscle tone. The investigators obtained many parameters like muscle stiffness, frequency and decrement.

CONTACTS AND LOCATIONS:
Overall Officials: Diego Serrano-Muñoz, MsC, Principal Investigator — Hospital Nacional de Parapléjicos de Toledo
Locations (1):
- Diego Serrano-Muñoz, Talavera de la Reina, Castille-La Mancha, Spain

IPD SHARING:
Plan to Share IPD: Yes